CLINICAL TRIAL: NCT03758040
Title: Mechanisms of Fall Resistance to Diverse Slipping Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0861-18-EP; 1R15AG063106 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-04

CONDITIONS: Slipping and Falls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slips on Turns (Experimental): Slips will be administered during walking on a curved paths of radii 1.0, or 2.0 meters in early, middle or late stance to the inside or outside foot.
  Interventions: Other: Slips on Turns
- Slips on Slopes (Experimental): Slips will be administered during walking on sloped ground of 5.0 or 10.0 degrees mediolaterally or anteroposteriorly, or flat ground, in early middle or late stance. For mediolateral slopes, slips will be administered to the uphill or downhill foot.
  Interventions: Other: Slips on Slopes

INTERVENTIONS:
Other: Slips on Turns — A slip will be administered to participants at 3 different times in the gait cycle for each of 3 different patch curvatures and 2 different legs for a total of 18 slip episodes. Slips will be delivered while walking along a straight path (infinite radius), or curved paths with radii 2, or 1 meters.
  Arms: Slips on Turns
Other: Slips on Slopes — Slips will be administered to participants at 3 different times in the gait cycle over sloped ground surface of no slope, ±5.0 and ±10.0 degrees slopes in the direction of walking, and 5.0 and 10.0 degrees perpendicular to the direction of walking. On slopes perpendicular to the direction of walking, slips will be administered to the uphill or downhill foot. A total of 27 slip episodes will be administered. Sloped walking surfaces will be generated with the Computer Assisted Rehabilitation Environment (CAREN) system treadmill.
  Arms: Slips on Slopes

SUMMARY:
Falls are the leading source of injury for all ages, and for older adults are the primary cause of injury related death. Loss of foot to ground traction accounts for 25-40% of falls, typically referred to as a slip. Slips alter the relationship between center of mass and lower limb base of support resulting in altered whole-body angular momentum and inability to support body weight due to loss of stability. But not all slips lead to falls. Stability may be recovered through a combination of response movements, such as swinging the arms or rapid recovery steps. Stability must be recovered quickly otherwise insufficient bodyweight support rapidly leads to a damaging ground collision. A high percentage of falls result in fractures, contusions and sprains to both the trunk and limbs, while slips disproportionately cause lower back injuries. A primary goal of fall prevention training is to improve the ability to resist slips using perturbations that mimic the specific sensory and biomechanical context of natural slip events. However, generating lifelike slip perturbations that mimic the diversity of slipping conditions poses a significant hurdle to improving a more general slip resistance ability. Using movement analysis, the investigators will determine the relationships between diverse slip conditions, reactive responses to slips from those conditions, and slip vulnerability across the gait cycle to generate new data that may guide future interventions.

DETAILED DESCRIPTION:
Recent evidence suggests most slip-related falls in daily life happen in diverse slipping conditions where the ground is not level, or the person is turning or changing direction. While slips that occur during straight walking on level ground and the responses to those slips are relatively well understood, very little is known about slips that occur while walking on slopes or curved paths and which reactive responses are effective to prevent falls in such conditions. This limits the ability of clinicians to incorporate a diverse range of slipping experiences into fall prevention interventions. Understanding how reactive responses and slip vulnerability depend on diverse slip conditions may guide future interventions that promote a more general fall resistance to the broader range of slips encountered in the real environment.

This project will determine the impact of turns and slopes on reactive movements and fall vulnerability by determining the effects of path curvature on reactive movements and slip vulnerability at different times in the gait cycle and determining the effects of ground slope on reactive movements and slip vulnerability at difference times in the gait cycle. It is hypothesized that diverse slipping conditions will change the reactive responses involving protective stepping and arm swing and that the distinct dynamics of turns and slopes produce maximum vulnerability to slips at different times in the gait cycle compared to slips during straight walking on level ground. To evaluate these aims, the investigators will administer slip perturbations on slopes that vary in both magnitude and direction, on curved paths that vary in curvature, and with slip onset that varies across early, middle, and late stance. Understanding the relationships between diverse slipping conditions, reactive responses, slip severity and fall vulnerability may guide future research and training interventions towards more comprehensive fall resistance ability.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-35

Exclusion Criteria:

* Uncontrolled hypertension
* Peripheral arterial disease
* Knee osteoarthritis
* Vertigo
* Meniere's disease
* Chronic dizziness
* History of back or lower extremity injury
* Surgery that affects mobility
* Neurological disease that limits the ability to walk

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel H Hunt, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Biomechanics Research Building, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests should be emailed to the PI.

RESULTS

PARTICIPANT FLOW:
Groups:
- Slips on Turns: Slips administered during walking on a straight path, or on curved paths of radii 1.0, or 2.0 meters in early, middle or late stance to the inside or outside foot.
  Slips on Turns: Subjects were administered a slip at 3 different times in the gait cycle for each of 3 different patch curvatures and 2 different legs for a total of 18 slip episodes. Slips were delivered while walking along a straight path (infinite radius), or curved paths with radii 2, or 1 meters.
- Slips on Slopes: Slips administered during walking on sloped ground of 5.0 or 10.0 degrees mediolaterally or anteroposteriorly, or flat ground, in early middle or late stance. For mediolateral slopes, slips were administered to the uphill or downhill foot.
  Slips on Slopes: Slips were administered at 3 different times in the gait cycle over sloped ground surface of no slope, ±5.0 and ±10.0 degrees slopes in the direction of walking, and 5.0 and 10.0 degrees perpendicular to the direction of walking. On slopes perpendicular to the direction of walking, slips will be administered to the uphill or downhill foot. A total of 27 slip episodes will be administered. Sloped walking surfaces will be generated with the Computer Assisted Rehabilitation Environment (CAREN) system treadmill.
Period: Overall Study
Arm/Group | Slips on Turns | Slips on Slopes
Started | 21 | 22
Completed | 21 | 21
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Slips on Slopes: Slips administered during walking on sloped ground of 5.0 or 10.0 degrees mediolaterally or anteroposteriorly, or flat ground, in early middle or late stance. For mediolateral slopes, slips were administered to the uphill or downhill foot.
  Slips on Slopes: Slips were administered at 3 different times in the gait cycle over sloped ground surface of no slope, ±5.0 and ±10.0 degrees slopes in the direction of walking, and 5.0 and 10.0 degrees perpendicular to the direction of walking. On slopes perpendicular to the direction of walking, slips will be administered to the uphill or downhill foot. A total of 27 slip episodes will be administered. Sloped walking surfaces will be generated with the CAREN system treadmill.
- Total: Total of all reporting groups
Arm/Group | Slips on Turns | Slips on Slopes | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 19 | 21 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 15 | 17 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: meters] | 1.72 (0.12) | 1.73 (0.08) | 1.72 (0.10)
Weight [Mean (Standard Deviation); unit: kilograms] | 71.72 (18.17) | 72.90 (12.80) | 72.36 (15.26)

OUTCOME MEASURES:

1. Primary Outcome: Fall Rates - Slips on Turns
Description: Percentage of trials which result in a fall is recorded. Falls are classified when a load cell embedded in the harness system measures support forces exceeding 30% body weight.
Time Frame: Up to 4 hours
Population: Subjects were administered a slip at 3 different times in the gait cycle for each of 3 different patch curvatures and 2 different legs for a total of 18 slip episodes. Slips were delivered while walking along a straight path (infinite radius), or curved paths with radii 2, or 1 meters.
Measure: Number; unit: Percent of trials resulting in falls.
Units Other Than Participants: Trials
Arm/Group | Slips on Turns
Number analyzed (Participants) | 21
Number analyzed (Trials) | 378
Percent of trials resulting in falls.
  Fall Rate, Straight Walking | 0
  Fall Rate, Curved Walking (2 meter radius), slip administered to the inside foot | 7.94
  Fall Rate, Curved Walking (2 meter radius), slip administered to the outside foot | 1.59
  Fall Rate, Curved Walking (1 meter radius), slip administered to the inside foot | 23.44
  Fall Rate, Curved Walking (1 meter radius), slip administered to the outside foot | 3.13

2. Primary Outcome: Fall Rates - Slips on Slopes
Description: as for outcome 1
Time Frame: Up to 4 hours
Population: Slips were administered at 3 different times in the gait cycle over sloped ground surface of no slope, ±5.0 and ±10.0 degrees slopes in the direction of walking, and 5.0 and 10.0 degrees perpendicular to the direction of walking. On slopes perpendicular to the direction of walking, slips will be administered to the uphill or downhill foot. A total of 27 slip episodes will be administered. Sloped walking surfaces will be generated with the CAREN system treadmill.
Measure: Number; unit: Percent of trials resulting in falls.
Units Other Than Participants: Trials
Arm/Group | Slips on Slopes
Number analyzed (Participants) | 21
Number analyzed (Trials) | 567
Percent of trials resulting in falls.
  Fall Rate, Level Walking | 6.35
  Fall Rate, Sloped Walking (5 degrees), Uphill Slope | 6.35
  Fall Rate, Sloped Walking (10 degrees), Uphill Slope | 50.79
  Fall Rate, Sloped Walking (5 degrees), Downhill Slope | 7.94
  Fall Rate, Sloped Walking (10 degrees), Downhill Slope | 44.44
  Fall Rate, Sloped Walking (5 degrees), Cross-Slope | 9.60
  Fall Rate, Sloped Walking (10 degrees), Cross-Slope | 44.00

3. Secondary Outcome: Slipping Foot Distance
Description: The distance travelled by the slipping foot relative to the center of mass following the administered slip perturbation
Time Frame: Up to 4 hours
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Slipping Foot Maximum Velocity
Description: The maximum velocity of the slipping foot relative to the center of mass following the administered slip perturbation
Time Frame: Up to 4 hours
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Trunk Maximum Angular Momentum
Description: The maximum angular momentum of the trunk following the administered slip perturbation
Time Frame: Up to 4 hours
Reporting Status: Not Posted, anticipated posting 2026-12

6. Secondary Outcome: Reactive Stepping Response Placement
Description: Position of the placement of the reactive stepping response relative to the center of mass following the administered slip perturbation
Time Frame: Up to 4 hours
Reporting Status: Not Posted, anticipated posting 2026-12

7. Secondary Outcome: Reactive Stepping Response Time
Description: Duration of time between the onset of the administered slip perturbation and the placement of the reactive stepping response
Time Frame: Up to 4 hours
Reporting Status: Not Posted, anticipated posting 2026-12

8. Secondary Outcome: Reactive Arm Swing Momentum Change
Description: The change in arm momentum between the onset of the administered slip perturbation and the end of the slip
Time Frame: Up to 4 hours
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: Up to 4 hours
Description: This protocol was not expected to put participants at risk for Serious Adverse Events, or at risk for All-Cause Mortality.
Arm/Group | Slips on Turns | Slips on Slopes
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

LIMITATIONS AND CAVEATS:
Fall rates for slipping on slopes are taken from walking trials on a treadmill. The moving treadmill belts require the participants to recover from the slip and continue walking. Therefore, the fall rates we measured are very likely to overestimate the fall rates from slips on slopes during walking overground.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT03758040/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT03758040/ICF_001.pdf